CLINICAL TRIAL: NCT04475107
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-Controlled, Phase Ⅱ Clinical Trial to Evaluate Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients
Brief Title: The Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-PA-COV-201
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: Pyramax; Pyronaridine; Artesunate; COVID-19; Corona virus
MeSH Terms: conditions — COVID-19 | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Pyramax (Pyronaridine 180mg/ Artesunate 60mg)
  Interventions: Drug: Pyronaridine-Artesunate
- Arm B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyronaridine-Artesunate — Pyramax
  Arms: Arm A
Drug: Placebo — Placebo
  Arms: Arm B

SUMMARY:
This study is a multi-center, randomized, double-blind, parallel, placebo-controlled, phase Ⅱ clinical trial to evaluate efficacy and safety of Pyramax in mild to moderate COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years at the time of signing Informed Consent Form
2. Body weight ≥45 kg at screening
3. Laboratory (rRT-PCR) confirmed infection with SARS-CoV-2 by testing specimens from upper airway (i.e. nasopharyngeal and oropharyngeal swab) or lower airway (i.e. sputum) within 96 hours of randomization
4. Oxygen saturation(SpO2) > 94% at randomization, in room air condition
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Diagnosed with severe pneumonia
2. Patients with clinically significant cardiovascular disease (including arrhythmia, QTc interval prolongation)
3. Patients with clinically significant anemia (Hemoglobin <8.0 g/dL)
4. Patient with known allergic reaction or contraindication to any of the investigational medicinal product (pyronaridine tetraphosphate, artesunate)
5. Patients with known history of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, etc.
6. Patients with the gastrointestinal disease and surgery to affect the absorption, distribution, metabolism and excretion of the drug, active gastritis, gastrointestinal tract / rectal bleeding, gastric ulcer, pancreatitis abnormalities (except simple appendectomy or hernia surgery)
7. Patients who received antiviral drugs that is intended to treat COVID-19, within 28 days prior to screening evaluation (can be enrolled into the study, if the patient has gone through a sufficient wash-out period)
8. Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2)
9. Patients with known severe liver disease (i.e. ALT or AST>5 times upper limit, nausea, abdominal pain associated with jaundice or Child-Pugh stage B or C)
10. Viral disease (HIV, HBV, HCV, etc.) other than COVID-19 that require administration of other antiviral agents
11. Patients that require ventilation therapy (e.g. non-invasive ventilation, invasive mechanical ventilation, extracorporeal membrane oxygenation, etc.)
12. Patients with chronic underlying disease (e.g. uncontrolled diabetes mellitus, chronic kidney disease, chronic liver disease, chronic pulmonary disease, chronic cardiovascular disease, blood cancer, cancer patients with cancer treatment, patients taking immunosuppressants), highly obese patients, dialysis patients, and transplant patients that are determined by the Physician, to be not suitable for trial involvement.
13. Pregnant or lactating women
14. Male or female of childbearing potential who has plans to become pregnant during the study period and for three months after the clinical study or who is not willing to take appropriate contraceptive measures

    *Hormonal contraception (contraceptive implant, injections, pills, etc.), IUDs, condoms (male) and contraceptive diaphragm or cap (female), sterilization (vasectomy, tubal ligation, etc.)
15. Participating in another clinical trial currently or within 28 days from signing the informed consent
16. Patients that are deemed ineligible to participate in the clinical trial by the Investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of patients with virological clearance of SARS-CoV-2 at day 7 post-dose* | Day 7
  * Patients who are rRT-PCR negative for COVID-19

SECONDARY OUTCOMES:
Viral load reduction of SARS-CoV-2 at Day 3, 7, 10, and 14 post-dose compared to the baseline | Day 3, 7, 10, 14
Proportion (%) of patients with virological clearance of SARS-CoV-2 at Day 3, 10, and 14 post-dose* | Day 3, 10, 14
  * Patients who are rRT-PCR negative for COVID-19
Change in WHO Ordinal Scale for Clinical Improvement at Day 3, 7, 10, 14, and 28 post-dose from the baseline | Day 3, 7, 10, 14, 28
Change in NEWS score at Day 3, 7, 10, 14, and 28 post-dose from the baseline | Day 3, 7, 10, 14, 28
Time to achieve normalization of body temperature, post-dose | Day 3, 7, 10, 14, 28
Time to achieve normalization of respiratory rate, post-dose | Day 3, 7, 10, 14, 28
Time to achieve normalization of oxygen saturation, post-dose | Day 3, 7, 10, 14, 28

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Korea University Ansan Hospital, Ansan
  - Chungnam national University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyungpook National University Hospital, Seoul
  - National Medical Center, Seoul
  - Sahmyook Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Marys' Hospital, Seoul
  - Ajou University Hospital, Suwon